CLINICAL TRIAL: NCT00312767
Title: A Multicenter, Open-Label, Cross-Over Trial to Evaluate the Pharmacokinetics of Fabrazyme During Simultaneous Fabrazyme Infusion and Chronic Hemodialysis in Patients With Fabry Disease.
Brief Title: A Study in Patients With Fabry Disease Who Are on Chronic Hemodialysis Therapy for Treatment of End-stage Renal Insufficiency.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Coporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AGAL03505
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Fabry Disease
Keywords: Agalsidase beta; alpha Galactosidase A; aGAL; rh aGAL; Fabry; GL3; Fabrazyme; dialysis; hemodialysis
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase beta

INTERVENTIONS:
Drug: Fabrazyme (agalsidase beta)

SUMMARY:
People with Fabry disease have an alteration in their genetic material (DNA) which causes a deficiency of the a-galactosidase A enzyme. Fabrazyme is a drug that helps to breakdown and remove certain types of fatty substances called "glycolipids." These glycolipids are normally present within the body in most cells. In Fabry disease, glycolipids build up in various tissues such as the liver, kidney, skin, and blood vessels because a-galactosidase A is not present, or is present in small quantities. The build up of glycolipid (globotriaosylceramide or GL-3) levels in these tissues in particular is thought to cause the clinical symptoms that are common to Fabry disease. This study is designed to verify that no loss of Fabrazyme occurs during simultaneous Fabrazyme infusion and hemodialysis in patients currently receiving Fabrazyme at a dose of 1.0 mg/kg every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient must provide signed, written informed consent prior to any study-related procedures being performed.
* Patient is between 18 and 65 years of age, inclusive.
* Patient has documented Fabry disease.
* Patient has received bi-weekly 1 mg/kg infusions of Fabrazyme for at least 6 months prior to enrollment into the study.
* Patient has not experienced moderate or severe infusion-associated reactions (IARs) from Fabrazyme infusions, which were also associated with a rate reduction, within 3 months prior to enrollment into the study.
* Patient has been receiving chronic hemodialysis for treatment of end-stage renal insufficiency for at least 3 months prior to enrollment into the study.
* Patient has good vascular access for hemodialysis.
* Patient has not and will not have any other (investigational) drug(s) infused during their hemodialysis, and is expected to have a stable concomitant medication regimen at all PK assessments.

Exclusion Criteria:

* Patient's hemoglobin is < 9 g/100 mL at Screening/Baseline.
* Patient has a clinically significant organic disease or an unstable condition that, in the opinion of the Investigator, would preclude participation in the study.
* Patient has a medical condition, serious intercurrent illness, or extenuating circumstance that would significantly decrease study compliance.
* Patient has participated in a study employing an investigational drug within 30 days prior to the start of their participation in this study.
* Patient is unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04

PRIMARY OUTCOMES:
Verify that no loss of Fabrazyme occurs during simultaneous Fabrazyme infusion and hemodialysis with a low-flux membrane.

SECONDARY OUTCOMES:
Verify that no loss of Fabrazyme occurs during simultaneous Fabrazyme infusion and hemodialysis with a high-flux membrane.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Trident Nephrology Associates, North Charleston, South Carolina, United States